CLINICAL TRIAL: NCT07010510
Title: Quality of Life in Operated Adult Patients With Tetralogy of Fallot and Correlation With Myocardial Strain Analysis by Cardiac Magnetic Resonance Imaging and Exercise Test
Brief Title: Quality of Life in Operated Adult Patients With Tetralogy of Fallot and Correlation With Myocardial Strain Analysis by CMR
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Abdelrahman Abdelgaber Abdelhafez, Doctor, Assiut University
Other Study IDs: QOL in TOF
Record Dates: First submitted 2025-05-27; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: TOF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with TOF: The study cohort consists of adult patients (≥18 years) with previously repaired Tetralogy of Fallot (TOF) who underwent routine clinical follow-up, including cardiac imaging, functional testing, and laboratory investigations. Patients included underwent surgical repair using either valve-sparing techniques or valved conduits and had follow-up assessments performed at least 3 months post-surgery. Data will be retrospectively collected from medical records, imaging databases, and clinical documentation. The cohort includes patients in sinus rhythm or with a documented history of ventricular arrhythmia, all of whom were referred for routine cardiovascular magnetic resonance (CMR) imaging and other functional assessments as part of standard care.
  Interventions: Diagnostic Test: CMR, stress ECG, Holter, BnP

INTERVENTIONS:
Diagnostic Test: CMR, stress ECG, Holter, BnP — This study involves no experimental intervention. All data were collected retrospectively from patients with repaired Tetralogy of Fallot (TOF) who underwent standard clinical follow-up. As part of routine care, patients received comprehensive multimodal functional assessment, including:
  Cardiac Magnetic Resonance Imaging (CMR) with feature-tracking strain analysis
  Transthoracic Echocardiography
  Exercise stress testing (treadmill ECG using Bruce protocol)
  12-lead ECG and 24-hour Holter monitoring
  Laboratory evaluation including NT-proBNP levels
  NYHA functional class assessment

SUMMARY:
Title:

Functional Assessment and Arrhythmia Prediction in Adult Patients with Repaired Tetralogy of Fallot Using a Multimodality Approach

Background:

Tetralogy of Fallot (TOF) is the most common cyanotic congenital heart defect. Surgical repair has improved survival into adulthood, but long-term complications like arrhythmias and heart failure remain common. Assessing health-related quality of life (HRQOL) and cardiac function is essential.

Aim:

Assess functional status of adult patients with repaired TOF using a multimodal approach, including myocardial strain analysis via CMR.

Identify predictors of arrhythmia using strain and clinical parameters.

Methods:

Design: Prospective observational study over one year.

Population: Adults (≥18 years) with repaired TOF undergoing follow-up CMR.

Assessments:

Clinical evaluation (NYHA class)

Echocardiography (RV size, function, valve status)

Laboratory tests (BNP, NT-proBNP)

Exercise testing (METs, VO₂ max)

ECG & 24-hour Holter monitoring (QRS duration, arrhythmias)

CMR (volumes, flow, fibrosis, strain analysis of RA, RV, LV)

Outcomes:

Primary: Functional assessment of repaired TOF patients.

Secondary: Detection of arrhythmia and need for further interventions (e.g., ICD or ablation).

Statistical Analysis:

Comparison between arrhythmic and non-arrhythmic groups.

Logistic regression for predictors of arrhythmia.

ROC analysis to determine optimal strain cut-off values.

Ethical Considerations:

Ethics committee approval and informed consent.

Data confidentiality maintained.

ELIGIBILITY:
* Inclusion criteria:

  * Adult TOF patients who were referred for surgical repair of TOF either valve sparing repair (VSR) or valved conduit (stented valve conduits, freestyle valved conduits, bio-prosthesis, or homograft).
  * Adults (age ≥18 years) with repaired TOF.
  * Undergoing routine CMR for clinical follow-up.
  * Sinus rhythm or known history of ventricular arrhythmia.
* Exclusion criteria:

  * Confounding other congenital defects e.g. AV canal.
  * Significant aortic regurgitation or stenosis.
  * Significant mitral regurgitation.
  * Residual significant major aorto-pulmonary collaterals (MAPCAs).
  * Patients with contraindications to CMR (e.g., pacemakers, severe renal impairment, claustrophobic).
  * Poor-quality CMR images precluding strain analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients (age ≥18 years) with previously repaired Tetralogy of Fallot (TOF), who were referred for routine clinical follow-up at least 3 months post-surgical correction. These patients underwent standard evaluations including cardiovascular magnetic resonance (CMR), transthoracic echocardiography, ECG, Holter monitoring, NT-proBNP measurement, and exercise stress testing. Patients were either in sinus rhythm or had a documented history of ventricular arrhythmia. Individuals with other major congenital heart defects, significant valvular disease, or contraindications to CMR were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
NYHA Class | 1 year
  New York Heart Association (NYHA) classification 1 to 4
cardiac magnetic resonance (CMR) | 1 years
  myocardial strain parameters
Exercise capacity (METs) | 1 years
  Functional capacity 1-15
NT-proBNP levels | 1 yeqrs
  Mg/dl

SECONDARY OUTCOMES:
Incidence of Arrhythmia in Adults with Repaired Tetralogy of Fallot (TOF) | At time of most recent follow-up (minimum 3 months post-surgical repair)
  Identification and documentation of arrhythmias based on standard 12-lead ECG and 24-hour Holter monitoring. Includes detection of premature ventricular contractions (PVCs), sustained or non-sustained ventricular tachycardia (VT), atrial flutter, atrial fibrillation, or other clinically significant arrhythmias requiring intervention.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Villafane J, Feinstein JA, Jenkins KJ, Vincent RN, Walsh EP, Dubin AM, Geva T, Towbin JA, Cohen MS, Fraser C, Dearani J, Rosenthal D, Kaufman B, Graham TP Jr; Adult Congenital and Pediatric Cardiology Section, American College of Cardiology. Hot topics in tetralogy of Fallot. J Am Coll Cardiol. 2013 Dec 10;62(23):2155-66. doi: 10.1016/j.jacc.2013.07.100. Epub 2013 Sep 27. PMID 24076489
- [Background] Carvalho JS, Shinebourne EA, Busst C, Rigby ML, Redington AN. Exercise capacity after complete repair of tetralogy of Fallot: deleterious effects of residual pulmonary regurgitation. Br Heart J. 1992 Jun;67(6):470-3. doi: 10.1136/hrt.67.6.470. PMID 1622697
- [Background] Steinmetz M, Stumpfig T, Seehase M, Schuster A, Kowallick J, Muller M, Unterberg-Buchwald C, Kutty S, Lotz J, Uecker M, Paul T. Impaired Exercise Tolerance in Repaired Tetralogy of Fallot Is Associated With Impaired Biventricular Contractile Reserve: An Exercise-Stress Real-Time Cardiovascular Magnetic Resonance Study. Circ Cardiovasc Imaging. 2021 Aug;14(8):e011823. doi: 10.1161/CIRCIMAGING.120.011823. Epub 2021 Aug 13. PMID 34384226
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Background] Baumgartner H, Hung J, Bermejo J, Chambers JB, Evangelista A, Griffin BP, Iung B, Otto CM, Pellikka PA, Quinones M; American Society of Echocardiography; European Association of Echocardiography. Echocardiographic assessment of valve stenosis: EAE/ASE recommendations for clinical practice. J Am Soc Echocardiogr. 2009 Jan;22(1):1-23; quiz 101-2. doi: 10.1016/j.echo.2008.11.029. No abstract available. PMID 19130998
- [Background] Renella P, Aboulhosn J, Lohan DG, Jonnala P, Finn JP, Satou GM, Williams RJ, Child JS. Two-dimensional and Doppler echocardiography reliably predict severe pulmonary regurgitation as quantified by cardiac magnetic resonance. J Am Soc Echocardiogr. 2010 Aug;23(8):880-6. doi: 10.1016/j.echo.2010.05.019. Epub 2010 Jul 1. PMID 20591618